CLINICAL TRIAL: NCT05117437
Title: The Effect Of Anaerobic Exercise On Bone Morphogenetic Protein 9
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Faruk Turgay, Associate Professor, Ege University
Other Study IDs: TDK-2020-22186; TDK-2020-22186 (Other Grant/Funding Number: Ege University Scientific Research Project Coordination Unit)
Record Dates: First submitted 2021-10-11; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Healthy; Exercise
Keywords: Bone morphogenetic protein; BMP9; anaerobic exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletic group: Healthy male athletes who have been doing regular anaerobic sports (such as basketball, volleyball and handball) for at least 3 months
  Interventions: Other: Physiological test; Other: Physical test; Other: Biochemical tests
- Control group: Healthy sedentary (not doing regular sports for at least 3 months) men with age and physical characteristics similar to the athlete group
  Interventions: Other: Physiological test; Other: Physical test; Other: Biochemical tests

INTERVENTIONS:
Other: Physiological test — This test was conducted to determine the endurance levels of the participants.
  Other Names: YOYO intermittent recovery test (level 1)
Other: Physical test — Height, weight, and BMI were determined
Other: Biochemical tests — BMP9, CTX1, COMP, oxLDL protein levels, ALP, GGT, TAS, TOS, OSI, NO, calcium, T-C, LDL-C, Triglyceride, HDL-C, glucose, CRP, AST, ALT, erythrocyte, mean erythrocyte volume (MCV), hematocrit, leukocyte, thrombocyte levels were determined from blood samples.

SUMMARY:
Bone morphogenetic protein (BMP) 9 from the BMP family has an important role in the remodeling of bone and cartilage. Due to these features, BMP9 can play an important role in especially anaerobic exercise training adaptations. However, the role of anaerobic exercise in these effects is still unclear. The aim of this study is to investigate the role of BMP9 on the effects of acute and chronic anaerobic exercise on bone metabolism markers. Postprandial venous blood samples were taken pre- and post- acute YOYO intermittent recovery test (level 1) in 40 trained male athletes aged 18-35 who did anaerobic sports (such as basketball, volleyball and handball) and 41 sedentary volunteers aged 18-35. Serum BMP9, as markers of bone formation and resorption; alkaline phosphatase (ALP), C-terminal telopeptide of type 1 collagen (CTX1), cartilage oligomeric matrix protein (COMP) and calcium levels were determined. The data to be obtained as a result of our study can give information about the relationship between the skeletal and bone health of the athletes and anaerobic exercise.

ELIGIBILITY:
Inclusion Criteria:

* being male
* having a body mass index of less than 30 being

Exclusion Criteria:

* to have some disease or disability
* to regularly use cigarettes and alcohol
* to use any medication or antioxidant substance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletic group: trained male athletes who did anaerobic sports (such as basketball, volleyball and handball) Control group: sedentary males
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from serum BMP9 levels at pre- and post- YOYO intermittent test | between 40-50 minutes
  Postprandial venous blood samples were obtained before and after acute YOYO IR test (level 1). The YOYO test lasted 10-20 minutes depending on the ability level of the participants. A blood sample was taken 15 minutes before and 15 minutes after the YOYO test. From these blood samples, serum Bone morphogenetic protein 9 (BMP9) was determined.
Change from serum CTX1 levels at pre- and post- YOYO intermittent test | between 40-50 minutes
  Postprandial venous blood samples were obtained before and after acute YOYO IR test (level 1). The YOYO test lasted 10-20 minutes depending on the ability level of the participants. A blood sample was taken 15 minutes before and 15 minutes after the YOYO test. From these blood samples, serum C-terminal telopeptide of Type 1 collagen (CTX1) was determined.
Change from serum COMP levels at pre- and post- YOYO intermittent test | between 40-50 minutes
  Postprandial venous blood samples were obtained before and after acute YOYO IR test (level 1). The YOYO test lasted 10-20 minutes depending on the ability level of the participants. A blood sample was taken 15 minutes before and 15 minutes after the YOYO test. From these blood samples, serum cartilage oligomeric matrix protein (COMP) was determined.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Turgay, Study Director — Ege University Faculty of Sport Sciences
Locations (1):
- Ege University Faculty of Sport Sciences, Izmir, Turkey (Türkiye)